CLINICAL TRIAL: NCT03777111
Title: Effect of Single and Double Task Training on Gait, Balance and Functional Mobility in the Elderly: Randomized Controlled Study
Brief Title: Effect of Single and Dual Task Training on Gait, Balance and Functional Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Emel TAŞVURAN HORATA, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 60116787-020/53283
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Aging
Keywords: Aging; gait; balance; functional mobility; dual task training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Task Training Group (Active Comparator): Gait and balance exercises will be applied in single task training group.
  * Semi-tandem, tandem stand with eyes open and close
  * One leg stance with eyes open and close
  * Gait exercises; walking forwards, backwards, sidewards, semi-tandem and tandem walking
  * Reaching forward and sidewards with eyes open and close
  Interventions: Other: Exercise
- Dual Task Training Group (Experimental): The exercises given in the single task training group will be combined with the cognitive tasks.
  * Semi-tandem, tandem stand with recall a sequence of numbers
  * One leg stance with writing pre-defined letters or words with other foot
  * Semi-tandem or tandem walking with saying previous number (one or two previous) from number that researcher has given before
  * Walking sidewards with collecting numbers that researcher has given
  * Walking backwards with counting forward by one (then two or three)
  * Reaching forward with counting backward one (then two or three)
  * Reaching sidewards with saying next number (one or two next) from number that researcher has given before
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Single Task Training: Single task training includes exercises that require only one task or stimulation. For this study the task consists of motor tasks (walking or balance) Dual Task Training: Dual task training includes exercises simultaneous performance of two tasks that can be performed independently, measured separately and with different goals. In the study motor tasks will combine with cognitive tasks.

SUMMARY:
Most of the daily life activities include dual task performance. Unlike conventional physiotherapy approaches, dual task training aims to improve both motor performance and cognitive performance at the same time. Geriatric rehabilitation approaches in Turkey; single task training (containing only motor performance) is applied to older adults for walking and balance disorders. Recent studies have shown gait parameters and balance abilities are influenced cognitive function and also dual task training is had to include in rehabilitation programs in order to improve walking and balance skills of the healthy elderly. In Turkey, a similar study is not found. The goal of this study is to evaluate in healthy elderly, effect of dual-task and single-task training on gait performance, and their effect on the balance abilities and functional mobility also to evaluate advantages one to another and to gain a different perspective to geriatric rehabilitation for the elderly in Turkey.

DETAILED DESCRIPTION:
Protocol:

In this study, the demographic information (age, gender, body mass index, education level, occupation, etc.) of all participants will be recorded first. In the first evaluation, the participants' gait parameters will be determined by using the 10-meter walking test and the wearable sensors. Balance is evaluated by Functional Reach Test, One Leg Stand Test and Tinetti Balance and Gait Assessment. Cognitive skills will be evaluated by using Mini Mental Test and Stroop Test. After the first evaluations of the participants, the participants will be given single or dual task training for 6 weeks, 2 times a week, not on consecutive days. If participants are absent for any training session, a compensation training session will be organized for them. After completing the single and / or dual task training, the final evaluations will be made. Randomization will be performed according to age, gender and body mass index of participants. After the randomization, participants' training group will be determined. Warm-up and cooling exercises will be carried out between 5-10 minutes before and after each training. Each training will consist of approximately 45-60 minutes including warm-up and cooling exercise periods. Each exercise starts with 5 repetitions and proceeds to 10 repetitions. To reduce the effects of fatigue and to draw attention, a break time that consists of approximately 1-2 minutes will be given.

Statistical Analysis:

The effect size obtained in the reference study was strong (d = 1.16). As a result of the power analysis using the effect size value in the reference study for the study, it was calculated that 80% power could be obtained at 95% confidence level when at least 20 people (10 people per group) were included the study. The data will be analyzed with Statistical Package for the Social Sciences (SPSS) package program. Continuous variables will be given as mean ± standard deviation and categorical variables as number and percentage. In the independent group comparisons, if the parametrical test assumptions are obtained, independent samples t-test will be used if the parametric test assumptions are not obtained Mann Whitney U test will be used. In the dependent group comparisons, when the parametric test assumptions are obtained, paired samples t-test; if not obtained Wilcoxon tests will be used.

ELIGIBILITY:
Inclusion Criteria:

* At least to graduate from primary school or ability to read and write
* Mini mental test score> 24
* Ability to achieve daily living activities independently
* Ability to walk independently in the community (at least 10 meters without walking aids)

Exclusion Criteria:

* Presence of acute (fracture, surgery), chronic (Parkinson's diseases, diabetes or stroke) and cognitive (Alzheimer, dementia, etc.) diseases
* Presence of hearing impairment that cannot be resolved by hearing devices and presence visual impairment that cannot be resolved by hearing aids.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
10 meter walk test | six week
  This test will perform with wearable gait sensors and will evaluate gait parameters.
Functional Reach Test | six week
  Balance test
One Leg stand Test | six week
  Balance test
Tinetti balance and gait assessment | six week
  For evaluating balance and gait
Stroop test | six week
  cognitive test

CONTACTS AND LOCATIONS:
Overall Officials: Suat EREL, Study Director — PhD
Locations (1):
- Pamukkale University, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shin SS, An DH. The Effect of Motor Dual-task Balance Training on Balance and Gait of Elderly Women. J Phys Ther Sci. 2014 Mar;26(3):359-61. doi: 10.1589/jpts.26.359. Epub 2014 Mar 25. PMID 24707083
- [Background] Brustio PR, Rabaglietti E, Formica S, Liubicich ME. Dual-task training in older adults: The effect of additional motor tasks on mobility performance. Arch Gerontol Geriatr. 2018 Mar-Apr;75:119-124. doi: 10.1016/j.archger.2017.12.003. Epub 2017 Dec 10. PMID 29245071
- [Derived] Tasvuran Horata E, Cetin SY, Erel S. Effects of individual progressive single- and dual-task training on gait and cognition among older healthy adults: a randomized-controlled comparison study. Eur Geriatr Med. 2021 Apr;12(2):363-370. doi: 10.1007/s41999-020-00429-5. Epub 2020 Nov 23. PMID 33226605